CLINICAL TRIAL: NCT07374146
Title: Research on the Individualized Treatment Strategy for Extremely Preterm Infants With hsPDA Based on Biomarkers and Targeted Delivery Systems
Acronym: BTDS-IT-hsPDA-
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Han Tongyan, attending doctor, Peking University Third Hospital
Other Study IDs: M20260024; A20260004 (Other: Peking university third hospital)
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hemodynamically Significant Patent Ductus Arteriosus
Keywords: Extremely premature infants; Biomarkers; Ibuprofen; Targeted delivery systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to address the need for individualized precision therapy for hemodynamically significant patent ductus arteriosus (hsPDA) in extremely preterm infants by integrating clinical biomarker screening with the design of a targeted drug-delivery system, and advancing early prediction and targeted intervention in a stepwise manner. Infants born at <32 weeks' gestational age will be enrolled. Multi-time-point blood samples and relevant clinical parameters will be systematically collected, with a focus on measuring cardiac function biomarkers (NT-proBNP), inflammatory cytokines (IL-6), angiogenic factors (VEGF), and hematologic indices (PCT and PLR). A multi-marker combined predictive model will be developed to improve the identification of high-risk infants. Building on this foundation, a nano-delivery system will be constructed via self-assembly of ibuprofen molecules and targeting ligands to achieve localized, precise, and controlled release at the ductus arteriosus. Its therapeutic efficacy and safety will be evaluated through in-vitro release testing, cytotoxicity assays, and animal model experiments.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32 weeks, regardless of sex;Parents or legal guardians are able to maintain effective communication with the investigators and agree to sign written informed consent.

Exclusion Criteria:

* Infants with severe congenital heart disease (other than PDA), such as severe tetralogy of Fallot, coarctation of the aorta, or pulmonary atresia;

Major structural malformations at birth, chromosomal abnormalities, or severe neurological defects;

Severe infection, bleeding tendency, or organ failure;

Contraindications to intravenous ibuprofen, including but not limited to: active gastrointestinal bleeding or a history of severe gastrointestinal bleeding; confirmed necrotizing enterocolitis or intestinal perforation; severe renal impairment (e.g., oliguria or elevated serum creatinine);

Prior treatment for PDA with other pharmacologic agents;

Deemed unsuitable for participation in this study by the treating physician.

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants (<32 weeks' gestation) receiving care at our hospital will be enrolled. Exclusion criteria include severe congenital heart disease other than PDA, major malformations, chromosomal abnormalities, severe neurologic defects, severe infection, bleeding tendency, organ failure, contraindications to intravenous ibuprofen, or prior pharmacologic PDA treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hsPDA | From birth until ductal closure or up to 3 weeks postnatal age
  Did hsPDA occur? (Yes/No)

SECONDARY OUTCOMES:
Trends in biomarker levels across different time points. | From birth until ductal closure or up to 3 weeks postnatal age